CLINICAL TRIAL: NCT04376996
Title: Slovenian National COVID-19 Prevalence Study
Acronym: SLO-COVID-19
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: ULMF2020-COVID-19
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and nasopharyngeal swab collected in Copan UTM media
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General cohort: General population cohort aged 0-100 years from Slovenia
  Interventions: Diagnostic Test: NO intervention planned due to the observational study design - only a diagnostic testing

INTERVENTIONS:
Diagnostic Test: NO intervention planned due to the observational study design - only a diagnostic testing — Only a diagnostic tests are planned: SARS-CoV-2 RNA in nasopharyngeal samples and anti-SARS-CoV-2 antibodies in blood

SUMMARY:
The investigators are conducting a national COVID-19 prevalence survey on a sample of 3,000 inhabitants that were randomly selected from the Slovenian population. The sample is representative in age, gender, and geographical distribution.

The main objective is to assess how many people in Slovenia have COVID-19 in April/May 2020 and how many were infected with SARS-CoV-2 previously.

The investigators are using a direct detection of SARS-CoV-2 RNA in nasopharyngeal samples with validated two-target PCR-based commercial assay. For a serological response to the etiological agent, IgG and IgA anti-SARS-CoV-2 antibodies are measured in plasma samples using a validated commercial assay.

DETAILED DESCRIPTION:
The investigators are conducting a national COVID-19 prevalence survey on a sample of 3,000 inhabitants that we have randomly selected from the Slovenian population. The sample is representative in age, gender, and geographical distribution.

The main objective is to assess how many people in Slovenia have COVID-19 in April/May 2020 and how many were infected with SARS-CoV-2 previously.

Direct detection of SARS-CoV-2 RNA in nasopharyngeal samples is performed with validated two-target PCR-based commercial assay. For a serological response to the etiological agent, IgG and IgA anti-SARS-CoV-2 antibodies are measured in plasma samples using a validated commercial assay.

Principal aims of the study are to systematically and accurately assess:

* How many people in Slovenia are actively infected with SARS CoV-2 in April/May 2020?
* How many are asymptomatic and do not even know they are or were infected?
* How many people in Slovenia have contacted SARS-CoV-2 and already have COVID-19 until mid May 2020?

The study is carried out by the Institute of Microbiology and Immunology of University of Ljubljana. The Institute is Slovenia's leading institution for microbiology and immunology research. The study is joined by a team of IT specialists, data scientists, and statisticians from the other departments of the University of Ljubljana.

To speed-up and support the study, an innovative information infrastructure for data gathering and management was purposely developed and optimized for the study. The system fosters error-free data collection, automatic processing of questionnaires using artificial intelligence approaches, and provides security for sensitive clinical data.

All participants will be passively followed up twice monthly and tested again for the presence of anti-SARS-CoV-2 antibodies in plasma samples six months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent only.

Exclusion Criteria:

Declined participation, no response on study invitation, no samples collected.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 3,000 inhabitants randomly selected from the Slovenian general population. Sample is representative in age, gender, and geographical distribution.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 RNA in nasopharyngeal samples | April to May 2020
  Prevalence of SARS-CoV-2 RNA in nasopharyngeal samples
Prevalence of anti-SARS-CoV-2 antibodies in blood samples | April to November 2020
  Prevalence of anti-SARS-CoV-2 antibodies in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Mario Poljak, MD, Principal Investigator — Univesity of Ljubljana, Slovenia
Locations (1):
- University of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maver Vodicar P, Ostrbenk Valencak A, Zupan B, Avsic Zupanc T, Kurdija S, Korva M, Petrovec M, Demsar J, Knap N, Strumbelj E, Vehovar V, Poljak M. Low prevalence of active COVID-19 in Slovenia: a nationwide population study of a probability-based sample. Clin Microbiol Infect. 2020 Nov;26(11):1514-1519. doi: 10.1016/j.cmi.2020.07.013. Epub 2020 Jul 18. PMID 32688068
- [Result] Poljak M, Ostrbenk Valencak A, Strumbelj E, Maver Vodicar P, Vehovar V, Resman Rus K, Korva M, Knap N, Seme K, Petrovec M, Zupan B, Demsar J, Kurdija S, Avsic Zupanc T. Seroprevalence of severe acute respiratory syndrome coronavirus 2 in Slovenia: results of two rounds of a nationwide population study on a probability-based sample, challenges and lessons learned. Clin Microbiol Infect. 2021 Jul;27(7):1039.e1-1039.e7. doi: 10.1016/j.cmi.2021.03.009. Epub 2021 Apr 7. PMID 33838303